CLINICAL TRIAL: NCT01781221
Title: Sinus Floor Elevation Using Separately Two Different Xenografts - A Prospective Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-200
Record Dates: First submitted 2013-01-10; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Posterior Maxilla Edentulous Patients With Insufficient Alveolar Bone Height

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Alpha-Bio's GRAFT Natural Bovine Bone (Active Comparator): two different bone substitutes commonly used in dental procedures.
  Interventions: Device: Alpha-Bio's GRAFT Natural Bovine Bone
- Bio-Oss xenograft (Active Comparator): two different bone substitutes commonly used in dental procedures.
  Interventions: Device: Bio-Oss xenograft

INTERVENTIONS:
Device: Alpha-Bio's GRAFT Natural Bovine Bone
  Arms: Alpha-Bio's GRAFT Natural Bovine Bone
Device: Bio-Oss xenograft
  Arms: Bio-Oss xenograft

SUMMARY:
The purpose of this study is to compare the regenerative results of using separately two different xenografts after two-step sinus floor elevation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will present with a moderately or severely atrophic posterior maxilla with 1-6 mm residual alveolar bone .
2. Men and women over the age of 18 years.
3. Patient has signed the Informed Consent.

Exclusion Criteria:

1. Chronic steroid therapy.
2. Uncontrolled diabetes.
3. Cardiovascular disease.
4. Past irradiation of head and neck.
5. Maxillary sinus cysts.
6. Active chronic sinusitis.
7. Smoking more than ten cigarettes per day during the 3 months preceding this study .
8. Malignant disease in the 5 years preceding this study.
9. Uncontrolled bleeding disorders such as: hemophilia, thrombocytopenia, granulocytopenia
10. Disease that compromise the immune system
11. Psychiatric disorder
12. Hypersensitivity to titanium, collagen or bovine bone.
13. Women who are pregnant or nursing.
14. Patients with non-treated periodontal disease.
15. Medical and/or general contraindications for intraoral surgical procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-02; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Uneventful healing and histological bone formation | 6 months following sinus floor augmentation

SECONDARY OUTCOMES:
X-ray demonstration of volume - stable results | 6 months following augmentation procedures.
Equally high implant survival rates and crestal bone loss | After 1,2 years